CLINICAL TRIAL: NCT02931682
Title: Observational Study of Males With Creatine Transporter Deficiency
Acronym: Vigilan
Status: Terminated | Type: Observational
Why Stopped: Sponsor decision not related to safety concerns
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: LUM-001-C-01; UX068-CL001 (Other: Ultragenyx Pharmaceutical Inc)
Record Dates: First submitted 2016-10-05; First posted 2016-10-13 (Estimated); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Creatine Deficiency, X-linked
Keywords: Creatine transporter; developmental delay; intellectual disability; X-linked; language; seizure; observational; brain spectroscopy
MeSH Terms: conditions — Creatine deficiency, X-linked; Learning Disabilities; Intellectual Disability; Language; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, cerebrospinal fluid, urine and fibroblasts
Oversight: Data Monitoring Committee: No

SUMMARY:
The objectives of this study are to illustrate the clinical, neuro/electrophysiologic, biochemical, and developmental status and progression of patients with Creatine Transporter Deficiency (CTD) and to evaluate the utility of performance-based and other measures in the CTD population.

DETAILED DESCRIPTION:
This is an observational study designed to determine an appropriate clinical assessment battery for males with CTD, and to evaluate Magnetic resonance spectroscopy (MRS) along with other potential biomarkers. It is designed to explore developmental domains of interest and to examine the feasibility and utility of various neuropsychological assessments to measure domains of interest, and to identify possible endpoints for interventional studies. Study will also explore genotype-phenotype correlations.

Clinical adverse events will be monitored throughout the study.

This study was previously posted by Lumos Pharma, which has been transferred to Ultragenyx in June 2019.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has genomic confirmation of a pathologic mutation in the SLC6A8 gene.
2. Subject is able to complete study-related procedures.
3. Subjects' parents/guardians/caregivers must provide written consent (informed consent) to study-related procedures, and if appropriate, the subject will provide an assent.

Exclusion Criteria:

1. Subject has had status epilepticus within 3 months of screening.
2. Subject is unable to comply with the study procedures or with a clinical disease or laboratory abnormality that in the opinion of the investigator would potentially increase the risk of participation.

Ages: 6 Months to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community Sample
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Change Over Time Through Month 48 in the Bayley Scales of Infant and Toddler Development, 4th Edition (Bayley-4) | Month 48

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Ultragenyx Pharmaceutical Inc
Locations (10):
- United States (9):
  - University of California San Diego, La Jolla, California
  - Rush University Medical Center, Chicago, Illinois
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller JS, Farmer C, Blair S, Bianconi S, Akshoomoff N, Anselm I, Barshop BA, Becker L, Bennett AE, Berry LN, Berry-Kravis EM, Bruchey A, Byars AW, Cimms T, Cecil KM, Covello M, Cubit LS, Das T, Davis RJ, Drye M, Ficicioglu C, Fulton JB, Goin-Kochel RP, Guthrie W, Hallinan BE, Hannah-Shmouni F, Gustafson KE, Koeberl DD, Longo N, Mamak E, Mercimek-Andrews S, Michalak C, Porter FD, Rahhal S, Rees L, Spiridigliozzi GA, Stone C, Sullivan NR, Sutton VR, Thomas RP, Udhnani M, Waisbren S, Xu M, Zhang L, Brandabur M, Thurm A. Longitudinal Characterization of Males With X-Linked Creatine Transporter Deficiency: Final Results of a Multiyear Observational Study. Pediatr Neurol. 2025 Oct 30;175:8-18. doi: 10.1016/j.pediatrneurol.2025.10.023. Online ahead of print. PMID 41260060
- [Derived] Campbell K, Cawley NX, Luke R, Scott KEJ, Johnson N, Farhat NY, Alexander D, Wassif CA, Li W, Cologna SM, Berry-Kravis E, Do AD, Dale RK, Porter FD. Identification of cerebral spinal fluid protein biomarkers in Niemann-Pick disease, type C1. Biomark Res. 2023 Jan 31;11(1):14. doi: 10.1186/s40364-023-00448-x. PMID 36721240